CLINICAL TRIAL: NCT00989794
Title: Phase I/II Study for the Safety and Performance of GELRIN C
Brief Title: Study to Evaluate the Safety and Performance of Treatment of Articular Cartilage Lesions Located on the Femoral Condyle With gelrinC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Regentis Biomaterials (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 004-00
Record Dates: First submitted 2009-10-04; First posted 2009-10-06 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Cartilage Lesion to the Femoral Condyle
Keywords: cartilage; implantation; chondrocyte; condyle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GelrinC (Experimental): GelrinC one step implantation to the femoral condyle lesion
  Interventions: Device: GelrinC

INTERVENTIONS:
Device: GelrinC — Applied once during surgery

SUMMARY:
This is a single arm, open label multi-center study to determine safety and the performance of the treatment of cartilage lesions located on the femoral condyle with GelrinC.

Patients meeting inclusion/exclusion criteria at screening will be enrolled into the study, and will receive treatment implantation into their cartilage lesions.

Treatment will consist of GelrinC implantations at the symptomatic lesion of femur rated as ICRS III, or IVA with less than 6 mm of bone loss below the subchondral plate.

The patients will undergo a rehabilitation program during the follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18 and 65 years of age.
2. Not more than two treatable symptomatic lesions which are NOT posterior; patient must present with pain in the index knee of moderate or severe level (VAS score ≥5)
3. If Female: Actively practicing a contraception method, or Practicing abstinence, or Surgically sterilized, or Postmenopausal
4. Understands and voluntarily signs and dates an informed consent document.
5. Grade 3 or 4 acute (traumatic) or chronic (degenerative) lesion
6. Willingness to follow standardized rehabilitation procedures.
7. Willingness and ability to comply with the requirements of this protocol, including returning for evaluation (clinical and imaging) at periodic intervals post-treatment.
8. Study knee has intact ligaments
9. Ipsilateral knee compartment has intact menisci (or requires partial meniscectomy resulting in stable menisci)
10. Contralateral knee is asymptomatic, stable and fully functional.
11. MRI obtained preoperatively within 3 months of Surgery

    Intraoperative Arthroscopic Confirmation:
12. one or two symptomatic lesions of the femur rated as ICRS III, or IVA with less than 6 mm of bone loss below the subchondral plate
13. Individual defect size between 1 cm2 - 6 cm2 after arthroscopic debridement

Exclusion Criteria:

1. More than two symptomatic lesions
2. Untreatable Posterior lesions
3. Lesion greater than 6cm2
4. ICRS Grade larger than grade II on a surface that directly opposes the defect
5. Osteoarthritis or avascular necrosis (clinical and/or radiographic diagnosis)
6. History of autoimmune disease or inflammatory arthropathy, such as rheumatoid arthritis, systemic lupus, active gout, septic or reactive arthritis including any history of a positive ANA blood test.
7. History of chronic debilitating systemic disease and any other unstable cardiac and pulmonary disorders.
8. History of current or prior malignancy within the last 5 years.
9. Patients treated in the affected knee with microfracture in the last 12m months or had prior tendon repair, meniscus repair, ligament repair or realignment surgery in the last 6 months.
10. Patient with prior total or subtotal meniscectomy.
11. Body Mass Index (BMI) >32 Kg/m2
12. 'Patients with known HIV, Hepatitis A, B, or C infections or other immunodeficient state.
13. Patients requiring immunosuppressive medications.
14. Clinically significant organic disease including clinically significant cardiovascular, pulmonary, neurologic, hepatic or renal disease or other medical condition, serious concurrent illness or extenuating circumstance that, in the opinion of the investigator, make the subject a poor candidate for participation in the study.
15. Patients received any other investigational products within 6 months prior to study enrollment.

17.Taking specific OA drugs such as chondroitin sulfate, diacerein, n-glucosamine, piascledine, capsaicin within 2 weeks of the screening 18.Is receiving prescription pain medication other than NSAIDs or acetaminophen for conditions unrelated to the index knee condition, chronic use of anticoagulant, or taking corticosteroids 19.Uncontrolled diabetes 20.Any concomitant painful or disabling disease of the spine, hips or lower limbs that would interfere with evaluation of the afflicted knee 21.Any clinically significant or symptomatic vascular or neurologic disorder of the lower extremities 22.Any evidence of the following diseases in the target joint : septic arthritis, inflammatory joint disease, gout, recurrent episodes of pseudogout, Paget's disease of bone, ochronosis, acromegaly, hemochromatosis, Wilson's disease, primary osteochondromatosis, heritable disorders, collagen gene mutation 23.Current diagnosis of osteomyelitis 24.Liver enzymes (SGOT, SGPT, Alkaline Phosphatase) of more than two times the upper limit of normal or any other result that is clinically important according to the Investigator 25.CRP > 10 mg/l 26.Clinically significant abnormal finding on screening laboratory parameters. 27.Clinically relevant compartment malalignment (> 5 degrees) as measured from the mechanical axis verified by clinical assessment or radiographic imaging when required 28.Patients with a history of bleeding disorders, patients receiving anti-platelet therapy or other anticoagulant medication use within 10 days prior to the beginning of the study, or patients in whom antiplatelet or other anticoagulant medication use is anticipated during the course of the study. However, patients on low-dose aspirin may be included in the study if aspirin therapy is interrupted at least 10 days before the treatment and not resumed until at least 2 weeks after the treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-09; Primary Completion 2015-12 (Actual); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
No device related AE, or SAE | 1 year
Improvement in KOOS over baseline | 18 months

SECONDARY OUTCOMES:
improvement in outcome based on questionnaires (KOOS, IKDC, VAS, SF-36) | 2 years
improvement in outcome based on MRI (MOCART) | 2 years

REFERENCES:
- [Derived] Schreiner MM, Raudner M, Szomolanyi P, Ohel K, Ben-Zur L, Juras V, Mlynarik V, Windhager R, Trattnig S. Chondral and Osteochondral Femoral Cartilage Lesions Treated with GelrinC: Significant Improvement of Radiological Outcome Over Time and Zonal Variation of the Repair Tissue Based on T2 Mapping at 24 Months. Cartilage. 2021 Dec;13(1_suppl):604S-616S. doi: 10.1177/1947603520926702. Epub 2020 Jun 4. PMID 32493044